CLINICAL TRIAL: NCT07042555
Title: Efficacy of Cognitive Behavior Therapy, Pelvic Floor Therapy and Pharmacotherapy in the Treatment of Chronic Pelvic Pain in Women: A Comparative Study
Brief Title: Efficacy of Cognitive Behavior Therapy for Treatment of Chronic Pelvic Pain in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Bushra Akram, PhD Scholar, Islamia University of Bahawalpur
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IslUB
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Chronic Pelvic Pain, Pelvic Pain, Women
MeSH Terms: conditions — Pelvic Pain | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cognitive Behavior Therapy for Chronic Pain (CBT-cp) (Experimental)
  Interventions: Behavioral: CBT-cp
- Pelvic Floor Therapy (PFT) (Experimental)
  Interventions: Other: Pelvic Floor Therapy
- Pharmacotherapy (Experimental)
  Interventions: Drug: Pharmacotherapy
- Integrated CBT-cp and PFT (Experimental)
  Interventions: Combination Product: CBT-cp+PFT
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: CBT-cp — The participants in CBT-cp arm will receive weekly sessions of Cognitive Behavior Therapy for Chronic Pain.
  Arms: Cognitive Behavior Therapy for Chronic Pain (CBT-cp)
Other: Pelvic Floor Therapy — The participants in PFT arm will receive weekly sessions of pelvic floor therapy.
  Arms: Pelvic Floor Therapy (PFT)
Drug: Pharmacotherapy — The participants in Pharmacotherapy arm will receive prescription and non prescription pain medication.
  Arms: Pharmacotherapy
Combination Product: CBT-cp+PFT — The participants in integrated arm will receive weekly sessions of both CBT-cp and PFT.
  Arms: Integrated CBT-cp and PFT
Other: Placebo — The participants in placebo arm will receive sham drug.
  Arms: Placebo

SUMMARY:
The study will employ 4 treatment arms and 1 placebo arm to compare efficacy of CBT, PFT, Pharmacotherapy, Integrated CBT and PFT modalities in the management of chronic pelvic pain in women.

ELIGIBILITY:
Inclusion Criteria:

Women of reproductive age, Women with CPP having no pathological or anatomical causes, Women with Overactive Bladder Syndrome Women with Vulvodynia.

Exclusion Criteria:

Women experiencing per-menopause or menopause, Women with medical, or gynecological or hormonal abnormalities, Women with mental disorders, Women who use substances.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ) | Up to 12 weeks

IPD SHARING:
Plan to Share IPD: Undecided